CLINICAL TRIAL: NCT00752427
Title: R076477-SCH-702: a 24 Week Open-Label Extension to R076477-SCH-302
Brief Title: 24-Week Open Label Extension to a Randomized, 6-Week Double Blind, Placebo Controlled Study, to Evaluate the Safety and Tolerability of Flexible Doses of Extended Release OROS® Paliperidone in the Treatment of Geriatric Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004423
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia: paliperidone
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Paliperidone ER OROS®

SUMMARY:
The purpose of this open-label study was to evaluate the safety and tolerability of flexible doses of Extended Release OROS® Paliperidone in the treatment of geriatric subjects with schizophrenia after completion of the initial double blind study

DETAILED DESCRIPTION:
The primary objective of the open-label extension phase was the long-term assessment of safety and tolerability of Extended Release (ER) OROS paliperidone (3 mg to 12 mg/day) in subjects (>65 years of age) with schizophrenia, and the secondary objective was the assessment of long-term efficacy.

Paliperidone ER OROS® tablet formulation (3 to 12 mg/day) to be taken orally

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had completed the double-blind phase or discontinued due to lack of efficacy after at least 21 days of treatment, who signed the informed consent for the open-label phase, and who the investigator agreed that open-label treatment was in the best interest of the subject were eligible to participate in the open label phase

Exclusion Criteria:

* Significant and/or unstable systemic illnesses
* Allergy or hypersensitivity to risperidone or paliperidone
* Significant risk of suicidal or violent behavior
* Biochemistry, hematology, or urinalysis results that are not within the laboratory's reference range, and that are deemed by the investigator to be clinically significant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-06; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Long-term assessment of safety and tolerability of Extended Release (ER) OROS paliperidone (3 mg to 12 mg/day) in subjects (>65 years of age) with schizophrenia

SECONDARY OUTCOMES:
Assessment of long-term efficacy of Extended Release (ER) OROS paliperidone (3 mg to 12 mg/day) in subjects (>65 years of age) with schizophrenia, .

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: 24-Week Open Label Extension to Evaluate the Safety and Tolerability of Flexible Doses of Extended Release OROS® Paliperidone in the Treatment of Geriatric Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=594&filename=CR004423_CSR.pdf